CLINICAL TRIAL: NCT06250335
Title: Impact of a Prebiotic Food-enriched Diet (PreFED) in Combination With Ipilimumab/Nivolumab Combination Immune Checkpoint Blockade (ICB) in ICB-refractory Melanoma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-1067; NCI-2024-01235 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: ICB-refractory Melanoma
MeSH Terms: interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients receive prebiotic food-enriched snacks and supportive nutritional counseling to increase prebiotic foods in diet.
  Interventions: Other: Prebiotic Food-Enriched Diet; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Other: Prebiotic Food-Enriched Diet — Given by PO
  Other Names: PreFED
Drug: Ipilimumab — Given by IV
Drug: Nivolumab — Given by IV

SUMMARY:
To learn about the possible effects of a prebiotic food-enriched diet (PreFED) targeting the gut microbiome in participants with ICI-refractory melanoma who are receiving the combination of ipilimumab and nivolumab as part of their standard care.

DETAILED DESCRIPTION:
Primary Objectives Determining the overall response rate (ORR) to PreFED intervention + Ipi/Nivo in ICB-refractory metastatic melanoma participants.

Secondary Objectives

1. Determine progression-free survival (PFS) and overall survival (OS) to PreFED + Ipi/Nivo in ICB refractory melanoma
2. Compliance and adherence to interventions
3. Determine the safety (AEs) and tolerability (GSRS-IBS) of the dietary intervention
4. Assess the rate of immune related adverse events in participants on immunotherapy receiving dietary interventions
5. Assess the effects of dietary intervention on systemic and tumor immunity
6. Assess the effect of dietary intervention on gut microbiome composition and networks
7. Assess the effects of dietary intervention on gut metabolic output and systemic metabolism
8. Assess the effects of dietary interventions on quality of life and other participant reported outcomes (PROs)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. English-speaking
3. Body mass index (BMI) 18.5-45 kg/m2
4. ECOG performance status of 0 or 1
5. Histologically confirmed stage III/IV, unresectable cutaneous melanoma. Asymptomatic brain metastases are allowed.
6. Prior treatment with anti-PD1 or anti-PD-1 + anti-LAG3 agents and documented disease progression either while on these agents or after stopping therapy without intervening therapy.
7. Planned initiation of standard-of-care Ipilimumab 3 mg/kg + Nivolumab 1 mg/kg
8. Measurable disease per RECIST 1.1
9. Self-reported willingness to eat the provided foods (with some tailoring to their food preferences)
10. Self-reported willingness to comply with scheduled visits, undergo venipuncture, provide stool samples.

Exclusion Criteria:

1. Prior treatment with anti-CTLA4
2. Mucosal or uveal melanoma
3. Concurrent malignancy requiring systemic therapy other than hormonal therapy.
4. History of inflammatory bowel disease, total colectomy, or bariatric surgery
5. Currently taking steroids > Prednisone 10 mg/day or equivalent
6. IV antibiotic use in the past month or oral antibiotic use in past 2 weeks
7. Regularly taking supplements containing prebiotics, fiber and/or probiotics, and unable/unwilling to discontinue for the purpose of the study.
8. Medical contraindications to the Intervention Diet as determined by the treating physician.
9. Self-reported major dietary restrictions, including but not limited to relevant food allergies, celiac disease, or diets such as vegan, ketogenic, extended fasting.
10. Insulin-dependent diabetes or conditions requiring bile-acid sequestrants.
11. Current smoker or heavy drinker (defined as >14 drinks per week) or current illicit drug use.
12. Currently pregnant, planning to become pregnant, or lactating.
13. Cognitively impaired adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-01-23 (Estimated); Study Completion 2029-01-23 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 2 years
  ORR is defined as the proportion of participants whose best overall response BOR is either CR or PR. Best overall response is defined as the best response designation recorded between the date of first dose and the date of first objectively documented progression or the date of subsequent therapy, whichever occurs first per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Baruch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org